CLINICAL TRIAL: NCT01521858
Title: Relations Between Hematologic Variables and Postoperative Bleeding in Total Hip Replacement Arthroplasty
Brief Title: THRA_hematologic Variables
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B_1111_140_103
Record Dates: First submitted 2012-01-09; First posted 2012-01-31 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Avascular Necrosis of Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Total hip replacement arthroplasty is a surgery having intra- and postoperative substantial blood loss. The investigators will investigate the relationship between the various hematologic variables and postoperative bleeding volume.

ELIGIBILITY:
Inclusion Criteria:

* avascular necrosis of hip
* total hip replacement arthroplasty

Exclusion Criteria:

* revision operation
* hematologic disease
* anticoagulant medication
* preoperative hemoglobin < 10 g/dl
* preoperative transfusion of red blood cells

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagosed with avascular necrosis of hip and undergoing total hip replacement arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
postoperative bleeding volume | at first postoperative day
Hemoglobin | preoperative 1 day and postoperative 1 day
hematocrit | preoperative 1 day and postoperative 1 day
platelet | preoperative 1 day and postoperative 1 day
prothrombin time_international normalized ratio | preoperative 1 day and postoperative 1 day
activated partial prothrombin time | preoperative 1 day and postoperative 1 day
fibrinogen concentration | preoperative 1 day and postoperative 1 day
Rotational thromboelastometry | preoperative 1 day and postoperative 1 day

SECONDARY OUTCOMES:
volume of infused fluid during operation | Period from starting to finishing the operation (During operaiton, an expected average of 3 hours)
  Infused total crystalloid and colloid volume during the operation will be recorded.
intraoperative urine output | Period from starting to finishing the operation (During operaiton, an expected average of 3 hours)
transfusion units | Period from starting to finishing the operation (During operaiton, an expected average of 3 hours) and postoperative first day
  Red blood cell

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea